CLINICAL TRIAL: NCT06651983
Title: Association of Inflammatory Factors With Complications in the Diabetic Population: a Cross-sectional Study
Status: Not yet recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2024-468
Record Dates: First submitted 2024-10-07; First posted 2024-10-22 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1.with complications 2.without complications: non-intervention

SUMMARY:
This study is a cross-sectional study of patients with diabetes. The main purpose of this study is to explore the relationship between inflammatory indicators, but not limited to inflammatory indicators, and diabetes complications, in order to find early predictors and screen out high-risk groups.

DETAILED DESCRIPTION:
Diabetes is one of the most important public health challenges of the 21st century, placing a heavy burden on societies and economies. The World Health Organization estimates that more than 10% of the world's population has diabetes or is at high risk of developing it. With the change of lifestyle, the number of people with diabetes is increasing, the types of complications are more and more complicated, and the time of complications is more and more earlier. Studies have found that the mechanism of diabetes has far exceeded the traditional mechanisms such as insulin resistance and glucose intolerance in the past, and the role of chronic low-grade inflammation in the whole course of diabetes should not be underestimated. At present, more and more researchers have explored the relationship between inflammation and certain clinical outcomes, such as diabetes, diabetes-related complications, hyperlipidemia, myocardial infarction, stroke, aneurysm, bladder cancer, etc.

The study found that people with diabetes had higher levels of inflammation than those without diabetes, with a statistically significant difference, and among people with diabetes, those with severe complications had higher levels of diabetes than those without complications, with a statistically significant difference. Jiachen Luo's study also confirmed that higher SII was associated with a poorer prognosis in patients with diabetes complicated by an acute myocardial infarction event. Nayili Mahemuti et al. 's analysis of NHANES found a positive association between SII and the risk of hyperlipidemia. Paul M Ridker also analyzed the participants in the PROMINENT, REDUCEIT and STRENGTH trials, which included participants who were taking statins and diagnosed with coronary atherosclerosis. CRP was found to be significantly associated with the occurrence of several adverse cardiovascular events (highest high-sensitive CRP quartile vs lowest high-sensitive CRP quartile, adjusted HR 1.31, 95% CI 1.20-1.43; P < 0.0001). The body is a complex and complex system, with glucose metabolism, lipid metabolism, inflammatory metabolism and other systems closely related. The physiological and pathological changes of diabetes stimulate the activation of chronic, low-grade and non-infectious inflammation in the body, while long-term inflammatory factors act on various tissues, organs and systems of the body, which in turn aggravate the occurrence and development of diabetes, making diabetes and inflammation cause and effect each other. On the basis of traditional inflammatory indicators, many new inflammatory indicators have been derived, and the relationship between these indicators and clinical outcomes has not been fully explored. It is of great significance to investigate the relationship between inflammation and diabetic complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a normative diagnosis of type 2 diabetes
* Age ≥20 years old, regardless of gender
* From January 2018 to August 2023, he was treated in Nanfang Hospital

Exclusion Criteria:

* In the acute infection phase
* The researchers judged that it was not suitable to participate in this study

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Diabetic patients with or without complications
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
C-reactive protein | In November-december 2024
  Data on inflammatory markers measured during hospitalization were collected in international units. C-reactive protein was measured and reported by the clinical laboratory of Nanfang Hospital under the condition of fasting.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology and Metabolism, Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No